CLINICAL TRIAL: NCT03728426
Title: A Phase 2 Study of Letermovir Treatment for Patients Experiencing Refractory or Resistant Cytomegalovirus Infection or Disease With Concurrent Organ Dysfunction
Brief Title: Letermovir Treatment for Refractory or Resistant Cytomegalovirus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amy C. Sherman, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Amy C. Sherman, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-348
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus Infections; CMV
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letermovir (Experimental): Open label letermovir will be administered daily for up to 12 weeks. The study allows an optional additional 12 weeks of treatment for secondary prophylaxis if clinically indicated.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Patients will receive intravenous or oral letermovir at a dose of 480mg/day.
  Patients weighing 40 or more kilograms will receive a second, loading, dose 12 hours after the first dose of letermovir treatment.
  For patients receiving concomitant cyclosporine treatment, the letermovir dose will be 240mg/day.
  Other Names: Prevymis

SUMMARY:
The trial will evaluate the safety and efficacy of letermovir antiviral treatment of active cytomegalovirus infection or cytomegalovirus disease in patients with infections that are refractory or resistant to available treatments or who are experiencing organ dysfunction that makes unsafe the use of available antiviral treatments.

DETAILED DESCRIPTION:
This is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved letermovir for treatment of cytomegalovirus infection, but it has approved letermovir for the prevention of cytomegalovirus infection in bone-marrow transplantation patients.

This is the first time that letermovir will be administered to children in a clinical trial.

Cytomegalovirus (CMV) is a common virus, which a majority of people acquire at some time in their life. CMV remains in your body, but does not cause symptoms in the majority of people. Patients with a weakened immune system (a system that protects you from infections) may be more at risk for the virus becoming active and causing damage to some of your organs, especially in the gut and lungs. If the virus becomes present above a certain quantity, the doctor usually prescribes a drug to treat the infection at this stage to avoid damage to the organs.

In this case, the virus is no longer responding to the prescribed drug, and other drug options will be harmful to the participant's health. Participants are being invited to take part in a research study for an investigational drug called letermovir. The purpose of this study is to find out whether letermovir is as effective and as safe in treating CMV infection in patients who cannot tolerate standard treatments such as ganciclovir or foscarnet.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years
* Weight ≥30 kg
* Transplant recipient (HCT, SOT) or other immunocompromised patients including those with HIV infection that require antiviral treatment for CMV.
* Documented CMV disease or persistent CMV infection (CMV virus load above 500 IU/mL on consecutive measurements, at least one day apart).
* CMV infection is refractory to treatment (defined as ≥14 days of standard CMV treatment without clinical improvement for CMV disease, or failure to achieve >1 log reduction in CMV VL after ≥14 days of standard treatment for CMV infection)16,17
* Current CMV infection has documented genotypic resistance to ganciclovir or foscarnet.
* For patients with any prior CMV infection episode that broke through letermovir prophylaxis, but not during the current CMV infection, documentation of letermovir susceptibility testing should demonstrate absence of letermovir mutations known to confer resistance to letermovir.
* Severe myelosuppression (ANC <1000/µL, Hemoglobin <8g/dL, or Platelets <25,000/µL)17 or renal dysfunction (estimated creatinine clearance <60 mL/min by MDRD in adults or < 60 ml/min/1.73 m2 by bedside Schwartz equation in < 18 years-old) at baseline or which develops during antiviral treatment.

  --Patients who develop severe myelosuppression or renal dysfunction during antiviral treatment as defined above are eligible without having to meet the refractoriness/antiviral resistance criterion.
* Combinations of genotypic antiviral resistance and organ dysfunction that lead to eligibility are presented in the full protocol eligibility table.
* The effects of letermovir on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of letermovir administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of letermovir administration.

  --Patients of childbearing potential must have a negative serum or urine pregnancy test.
* Able to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to letermovir.
* Known history of cirrhosis with Child-Pugh Class C hepatic insufficiency at screening.
* Acute liver injury at baseline meeting Hy's law.
* Current CMV infection broke through letermovir prophylaxis.
* Patients with life expectancy of less than a week. Determination of life expectancy will be discussed with the patient's primary treatment physician.
* Patient taking strong inhibitors or inducers of hepatic CYP enzymes including rifampicin, phenytoin, clarithromycin, ritonavir, or cobicistat.
* HIV patients who are receiving antiretroviral treatment protease inhibitors (darunavir, lopinavir, etc) whether by themselves or boosted with ritonavir or cobicistat, or HIV patients receiving cyclosporine treatment due to strong drug-drug interactions.
* Combinations of genotypic antiviral resistance and organ dysfunction that do not meet eligibility criteria are described in the full protocol eligibility table.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Sherman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658
- [Derived] Imlay HN, Kaul DR. Letermovir and Maribavir for the Treatment and Prevention of Cytomegalovirus Infection in Solid Organ and Stem Cell Transplant Recipients. Clin Infect Dis. 2021 Jul 1;73(1):156-160. doi: 10.1093/cid/ciaa1713. PMID 33197929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 163 individuals were screened, 10 were enrolled in the study from Dana-Farber Cancer Institute inpatient and outpatient settings.
Groups:
- Letermovir: Open label letermovir will be administered daily for up to 12 weeks. The study allows an optional additional 12 weeks of treatment for secondary prophylaxis if clinically indicated.
  Letermovir: Patients will receive intravenous or oral letermovir at a dose of 480mg/day.
  Patients weighing 40 or more kilograms will receive a second, loading, dose 12 hours after the first dose of letermovir treatment.
  For patients receiving concomitant cyclosporine treatment, the letermovir dose will be 240mg/day.
Period: Overall Study
Arm/Group | Letermovir
Started | 10
Completed | 7
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Letermovir
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.15 [56.32 to 69.87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline CMV viral load [Median (Inter-Quartile Range); unit: IU/mL] | 1272 [925 to 2546]

OUTCOME MEASURES:

1. Primary Outcome: Virological Response on Treatment Week 6
Description: The virologic response milestones are defined as: 1) Any decrease in CMV DNA from baseline (Week 0), measured on week 3 and 2) A ≥2 log decrease in CMV DNA from baseline, or an undetectable CMV DNA, measured on week 6.
  For patients with clinical CMV disease, the clinical response milestones are defined as: 1) Stabilization of clinical disease by week 3 (i.e. no worsening signs or symptoms compared to week 1) as assessed by the site investigator and 2) Improvement or resolution of clinical disease by week 6 (i.e., improvement in signs and symptoms of affected organs [resolution of diarrhea, pneumonia, hepatitis, retinitis, etc.]) 3) Patients with clinical CMV disease should also meet virological response milestones outlined above to support the continuation of letermovir therapy. Patients who enter the study based solely on documented CMV disease by histopathology in the absence of quantifiable CMV virus load should remain nonquantifiable (less than 137 IU/mL).
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 10
Participants | 5

2. Secondary Outcome: Overall Survival
Description: number of patients alive
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 10
Participants | 7

3. Secondary Outcome: CMV Progression-free Survival
Description: Time from study enrollment to CMV progression or death whichever occurs first
Time Frame: 6 months
Population: 5 participants had CMV progression or death
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Letermovir
Number analyzed (Participants) | 5
days | 13 [13 to 19]

4. Secondary Outcome: Kinetics of Viral Clearance
Description: time to undetectable plasma CMV DNA
Time Frame: 6 months
Population: All participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Letermovir
Number analyzed (Participants) | 10
days | 166 [147 to 168]

5. Secondary Outcome: Percent of Patients With a Clinically Meaningful Treatment Response to Letermovir Treatment
Description: Virological response and a concomitant clinical response in patients with CMV disease by Week 6 of treatment.
  For patients with clinical CMV disease, the clinical response milestones are defined as:
  1. Stabilization of clinical disease by week 3 (i.e. no worsening signs or symptoms compared to week 1) as assessed by the site investigator and
  2. Improvement or resolution of clinical disease by week 6 (i.e., improvement in signs and symptoms of affected organs [resolution of diarrhea, pneumonia, hepatitis, retinitis, etc.])
  3. Patients with clinical CMV disease should also meet virological response milestones outlined above to support the continuation of letermovir therapy. Patients who enter the study based solely on documented CMV disease by histopathology in the absence of quantifiable CMV virus load should remain nonquantifiable (less than 137 IU/mL).
Time Frame: 6 Weeks
Population: 1 participant met the definition for CMV disease
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Emergence of Letermovir-resistant CMV Virus in Patients Treated in This Setting
Description: Number of participants with breakthrough letermovir-resistant CMV infection in patients receiving letermovir treatment who experienced an initial virological response.
Time Frame: 6 months
Population: All participants analyzed for letermovir breakthrough infections
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definitions aligned with clinicaltrials.gov definitions.
  All Adverse Events must be reported in routine study data submissions to the Overall PI on the toxicity case report forms. Investigators must report any adverse event (AE) that occurs after the initial dose of study treatment, during treatment, or within 30 days of the last dose of treatment on the local institutional SAE form.
Groups:
- Letermovir: Open label letermovir will be administered daily for up to 12 weeks. The study allows an optional additional 12 weeks of treatment for secondary prophylaxis if clinically indicated.
  Letermovir: Patients will receive intravenous or oral letermovir at a dose of 480mg/day.
  8 participants received the dose of 480mg/day, and 2 participants receiving cyclosporine received 240mg/day, which is the standard adjusted dose based on well-known interactions between letermovir and cyclosporine. Based on prior pharmacokinetic studies of letermovir, no adverse events related to the dose used for dose-adjustment are expected.
Arm/Group | Letermovir
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letermovir (N=10)
Diarrhea (Gastrointestinal disorders) | 1
Lung Infection (Infections and infestations) | 2
Heart Failure (Cardiac disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1 — Worsening refractory acute graft versus host disease
Cardiac Arrest (Cardiac disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letermovir (N=10)
Nausea (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 2
Bacteremia (Infections and infestations) | 2
Epistaxis (Blood and lymphatic system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Vascular disorders (Vascular disorders) | 2 — 1 participant with multiple ecchymoses, 1 participant with petechiae on left hand
Acidosis (Metabolism and nutrition disorders) | 1
Alkaline phosphatase increased (Hepatobiliary disorders) | 1
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1
Bone infection (Infections and infestations) | 1
Bruising (Blood and lymphatic system disorders) | 1
Disease progression of hematologic malignancy (Blood and lymphatic system disorders) | 1
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 — Ear fullness
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 1 — upper GI bleed
Headache (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 1 — Liver graft v host disease
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Infections and infestations (Infections and infestations) | 1 — Recurrent CMV viremia
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 — Laceration of back
Insomnia (General disorders) | 1
Malaise (General disorders) | 1
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
peripheral ischemia (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 — scab in left buttocks
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Vertigo (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Increased monocytes (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
This study did not reach the target number of participants needed to achieve target power and statistically reliable results. The study was closed early due to difficulty in recruiting during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03728426/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT03728426/ICF_002.pdf